CLINICAL TRIAL: NCT00699049
Title: A Randomized, Double Blind, Placebo-Controlled, Parallel Group Comparison of the Efficacy and Safety of Any Alpha Blocker Monotherapy and Any Alpha Blocker Plus Solifenacin in Men With Residual Overactive Bladder Symptoms of Urinary Frequency and Urgency With/Without Urgency Incontinence After Previous Monotherapy With Any Alpha Blocker
Brief Title: A Study Comparing the Efficacy of an Alpha Blocker Versus an Alpha Blocker Plus Solifenacin in Men With Overactive Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KYU-SUNG LEE (Other)
Collaborators: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor-Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMK-1
Record Dates: First submitted 2008-06-16; First posted 2008-06-17 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Urinary Bladder, Overactive
Keywords: Alpha blocker; Tamsulosin; Solifenacin; Overactive Bladder; Urgency incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Adrenergic alpha-Antagonists; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alpha blocker and placebo (Placebo Comparator)
  Interventions: Drug: Alpha blocker; Drug: placebo
- Alpha blocker and solifenacin (Experimental)
  Interventions: Drug: Alpha blocker; Drug: solifenacin

INTERVENTIONS:
Drug: Alpha blocker — oral
Drug: placebo — oral
  Arms: Alpha blocker and placebo
Drug: solifenacin — oral
  Other Names: Vesicare; YM905
  Arms: Alpha blocker and solifenacin

SUMMARY:
The purpose of this study is to explore additional benefit of solifenacin after 12-week treatment, compared with alpha blocker monotherapy in men with residual OAB symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Persistent symptoms of OAB as verified by the 3 day voiding diary, defined by:

  * symptoms of urinary urgency (defined as a level of >=3 in a 5 point urgency scale) at least two episode per 24 hours and
  * symptoms of urinary frequency ( >8 micturitions per 24 hours)
* On a stable dose of tamsulosin for at least 1 month

Exclusion Criteria:

* Previous history of acute urinary retention
* Patients have a baseline post-void residual (PVR) which exceeded 50% of voided urine volume
* Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
* Symptomatic acute urinary tract infection (UTI) during the screening period
* Treatment within the 14 days preceding randomization, or expected to initiate treatment during the study with any anticholinergic drugs and drug treatment for overactive bladder
* A 5-alpha reductase inhibitor if started less than 3 months prior to screening
* Patients with previous urethral, prostate or bladder neck surgery

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2008-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Achievement level of patients' individual satisfaction | At weeks 4 and 12

SECONDARY OUTCOMES:
Changes in urgency episodes | At weeks 4 and 12
Changes in OAB symptom scores | At weeks 4 and 12
Changes in QoL score by OAB-q | At weeks 4 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (3):
- South Korea (3):
  - Cheonan
  - Pusan
  - Seoul